CLINICAL TRIAL: NCT03094377
Title: Effect of Multisensory Stimulation on Upper Extremity Motor Recovery in Stroke Patient: a Preliminary Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Ray KF Li, Principal Investigator, Adjunct Lecturer, Tung Wah College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1193-6547
Record Dates: First submitted 2017-03-13; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Stroke
Keywords: Multisensory stimulation; motor recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This was a quasi-randomized-controlled pilot. Participants were randomly allocated by admission sequence to a multisensory therapy group or a conventional training group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensory therapy group (Experimental): The Multisensory therapy (MT) group received a 12-weeks (two sessions/ week; 90 minutes/session) training conducted by an occupational therapist. Each session began with 15 minutes of sensory stimulation (cold and vibration), 45 minutes of motor training and 30 minutes of self-care training.
  Interventions: Other: Multisensory therapy
- Conventional training group (Active Comparator): The conventional training (CT) group included 12 weeks (two sessions/ week; 90 minutes/session) training conducted by an occupational therapist. Each session included 60 minutes of upper extremity motor practice (same as in MT group) and 30 minutes of self-care training (same as in MT group).
  Interventions: Other: Conventional training

INTERVENTIONS:
Other: Multisensory therapy — Sensory stimulation, motor training and ADL training
  Arms: Multisensory therapy group
Other: Conventional training — Motor training and ADL training
  Arms: Conventional training group

SUMMARY:
Despite the advances in stroke rehabilitation, post-stroke upper extremity impairment is still a major challenge. Increasing evidence can be found supporting stimulation of the afferent receptor enhances neuroplasticity in the brain. Studies have suggested multisensory stimulation could promote motor learning by re-establishing the disrupted sensorimotor loop due to stroke and enhance neuroplasticity.

The objective of the study was to examine the effect of multisensory stimulation on upper-extremity motor recovery and self-care function in stroke patients.

DETAILED DESCRIPTION:
Stroke patients referred to occupational therapy division of geriatric day hospital will be recruited and randomly assigned to a multisensory therapy group or a conventional training group. The Multisensory therapy group received 12 weeks (two sessions/ week; 90 minutes/session) training. Each session began with 15 minutes of sensory stimulation (cold and vibration), 45 minutes of motor training and 30 minutes of self-care training. The conventional training group included 12 weeks (two sessions/ week; 90 minutes/session) training. Each session included 60 minutes of upper extremity motor practice and 30 minutes of self-care training.

Outcome measures included: Brunnstrom's stage, Fugl-Meyer Assessment Scale and Functional Test for the Hemiplegic Upper Extremity were used for upper limb motor control and function; and Manual muscle testing was used for muscle strength. The modified Barthel Index was used for self-care performance

ELIGIBILITY:
Inclusion criteria:

* First-time ischemic or hemorrhagic stroke;
* Stroke onset > 4 weeks and < 6 months
* Single lesion
* Upper extremity motor deficit
* No severe cognitive impairment and able to follow verbal instructions.

Exclusion Criteria:

* Skin conditions/ injuries over the stimulation application areas
* Contraindication for cold or vibration application
* Speech disorder or global aphasia
* Musculoskeletal or cardiac disorders
* Other neurological conditions
* History of diabetes or sensory impairment attributable to peripheral vascular disease or neuropathy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Fugl-Meyer Assessment of Motor Recovery at 3 months | Baseline and post intervention at week 12
  The Fugl-Meyer Assessment was used to assess the progress in synergistic and voluntary movement at baseline and post intervention.
Change from baseline Functional Test for the Hemiplegic Upper Extremity at 3 months | Baseline and post intervention at week 12
  The Functional Test for the Hemiplegic Upper Extremity was used to evaluate the recovery of the hemiplegic upper extremity functions at baseline and post intervention.

SECONDARY OUTCOMES:
Change from baseline Modified Barthel Index at 3 months | Baseline and post intervention at week 12
  The Modified Barthel Index was used to measure functional performance in basic activities of daily living at baseline and post intervention.
Change from baseline Manual Muscle testing at 3 months | Baseline and post intervention at week 12
  Manual muscle testing (MMT) was used for the evaluation of the motor recovery and strength of upper extremity muscle groups at baseline and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ray Li, Master, Principal Investigator — Occupational Therapist
Locations (1):
- Wong Tai Sin Hospital, Wong Tai Sin, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Share all the available data as requested